CLINICAL TRIAL: NCT05398731
Title: Risk of COVID 19 Disease Among Hypertensive Patients Using Angiotensin Converting Enzyme Inhibitors or Angiotensin Receptor Blockers At Assiut University Hospitals
Brief Title: Angiotensin Converting Enzyme Inhibitors and Angiotensin Receptor Blockers With Risk of COVID_19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Mohamed Abd Alwahab Abd Alhafz, Resident doctor, Assiut University
Other Study IDs: ACEI,ARBS and risk of COVID_19
Record Dates: First submitted 2022-05-19; First posted 2022-06-01 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients received ACEI: patient who use ACEI ( Duration, type of response, and the time period between the begining of and the emergence of symptoms of COVID-19)
  Interventions: Other: Covid_19
- patients received ARBs: patient who use ARBs ( Duration, type of response, and the time period between the begining of and the emergence of symptoms of COVID-19)
  Interventions: Other: Covid_19
- other antihypertensive drugs: patient who use other antihypertensive drugs(for example ca channel blockers and Beta blockers) ( Duration, type of response, and the time period between the begining of and the emergence of symptoms of COVID-19)
  Interventions: Other: Covid_19
- non hypertensive group: Non hypertensive persons with matched age and sex
  Interventions: Other: Covid_19

INTERVENTIONS:
Other: Covid_19 — Duration, type of response, and the time period between the begining of drug and the emergence of symptoms of COVID-19
  Other Names: ARBs; ca channel blockers; Beta blockers

SUMMARY:
1. To determine the risk of COVID -19 in patients who use ACEI and ARBS
2. To determine the Effect of ACEI and ARBS on COVID -19 infection .
3. To determine the Severity of COVID -19 in patients who use ACEI and ARBS .

DETAILED DESCRIPTION:
SARS -CORONA VIRUS -2 (COVID-19 disease) is an infectious disease caused by the SARS-CoV-2 virus The virus enters the body through the nose, eyes, or mouth. The spike protein binds specifically to the ACE2 receptors present on the type 2 pneumocytes in the alveoli in the lungs . (Fehr and Perlman, 2015) The binding of the ACE2 receptor allows the entry of the virus into the host cell .

The virus enters the host cell either by direct cell entry by membrane fusion or by endocytosis .(Wang , et al. 2008).

ACE inhibitors (angiotensin converting enzyme inhibitors) work by preventing angiotensin I from converting into angiotensin II. (Byrd,et al. 2019)

ARBs (Angiotensin receptor blockers)reduce the action of the hormone angiotensin II, by blocking receptors that the hormone acts on, specifically AT1 receptors, which are found in the heart, blood vessels and kidneys. (Byrd,et al. 2019) ACE inhibitors and ARBs are used to treat high blood pressure and congestive heart failure, to prevent kidney failure in patients with high blood pressure or diabetes, and to reduce the risk of stroke. (Byrd,et al. 2019) Continued use of ACEI/ARB has become controversial in the setting of COVID-19. The reason for this controversy stems from the fact that ACEIs and ARBs use may increase the expression of ACE2 receptor in animal-based studies, which is the known cellular receptor and a necessary entry point for SARS-COV-2 infection, as it has been indicated that ACE2 expression is downregulated following SARS infection, resulting in excessive activation of RAS and exacerbated pneumonia progression.(Peng Zhang.et al.april2020) It has rather been suggested that despite increasing ACE2 levels, ACE inhibitors and ARBs may rather play a protective role. ACEI, by reducing the conversion of angiotensin I (ATI) to angiotensin II (ATII) and ARBs, by reducing the binding of ATII to angiotensin I receptor may tilt the scale suggested by Bombardini et al. in favour of a protective ACE2-signalling pathway .( Bombardini T, Picano E.2020).

Reynolds et.al (2020)found no association between ACE inhibitors and ARBs and increase likelihood of a positive test for covid- 19 or its severity. (Reynolds et.al (2020) However, due to lack of sufficient clinical data supporting either the beneficial or harmful effects of ACEI/ARBs use in patients with COVID-19, the optimal strategy for the management of hypertension in COVID-19 is uncertain and remains to be elucidated. So The aim of this observational study was to determine the association between hypertensive patients using ACEI/ARBs and morbidity and mortality of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* patients who use ACEI
* patients who use ARBs
* patients who use other antihypertensive drugs(for example ca channel blockers or Beta blockers)
* Non hypertensive persons with matched age and sex

Exclusion Criteria:

1. < 18 years old.
2. Pregnant or breast-feeding patients.
3. Patients with autoimmune disease.
4. Patients with multi organ failure, active cancer, renal insufficiency or chronic kidney disease.
5. Patients received immunosuppressive drugs.
6. Immune compromised patients.
7. Patients with obstructive lung disease

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: questionnaire with 5 Domain:
  1. Personal and demographic data, socioeconomic status. and other co comorbid diseases.
  2. Included patients(groups)
  3. Adherence of the patients to precautions against SARS-COV2.
  4. SARS-CoV-2 infection:
  5. Post COVID- 19 symptoms.
  6. any investigation with the pt
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
determine the risk of COVID -19 in patients who use ACEI and ARBS | from begining of Covid_19 pandemic up till now
  determine the risk of COVID -19 in patients who use ACEI and ARBS

SECONDARY OUTCOMES:
determine the morbidity and Severity of COVID -19 in patients who use ACEI and ARBS | from begining of Covid_19 pandemic up till now
  determine the morbidity and Severity of COVID -19 in patients who use ACEI and ARBS

CONTACTS AND LOCATIONS:
Overall Officials: Hanan M Adawy Nafeh, PhD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Fehr AR, Perlman S. Coronaviruses: an overview of their replication and pathogenesis. Methods Mol Biol. 2015;1282:1-23. doi: 10.1007/978-1-4939-2438-7_1. PMID 25720466
- [Background] Wang H, Yang P, Liu K, Guo F, Zhang Y, Zhang G, Jiang C. SARS coronavirus entry into host cells through a novel clathrin- and caveolae-independent endocytic pathway. Cell Res. 2008 Feb;18(2):290-301. doi: 10.1038/cr.2008.15. PMID 18227861
- [Background] Byrd, James Brian; Ram, C. Venkata S.; Lerma, Edgar V. 2019
- [Background] Peng Zhang, Lihua Zhu, Jingjing Cai, Fang Lei, Juan-Juan Qin, Jing Xie, Ye-Mao Liu, Yan-Ci Zhao, Xuewei Huang, Lijin Lin, Meng Xia, Ming-Ming Chen, Xu Cheng, Xiao Zhang, Deliang Guo, Yuanyuan Peng, Yan-Xiao Ji, Jing Chen, Zhi-Gang She, Yibin Wang, Qingbo Xu, Renfu Tan, Haitao Wang, Jun Lin, Pengcheng Luo, Shouzhi Fu, Hongbin Cai, Ping Ye, Bing Xiao, Weiming Mao, Liming Liu, Youqin Yan, Mingyu Liu, Manhua Chen, Xiao-Jing Zhang, Xinghuan Wang, Rhian M. Touyz, Jiahong Xia, Bing-Hong Zhang, Xiaodong Huang, Yufeng Yuan, Rohit Loomba, Peter P. Liu, and Hongliang Li.April 2020
- [Background] Bombardini T, Picano E. Angiotensin-Converting Enzyme 2 as the Molecular Bridge Between Epidemiologic and Clinical Features of COVID-19. Can J Cardiol. 2020 May;36(5):784.e1-784.e2. doi: 10.1016/j.cjca.2020.03.026. Epub 2020 Mar 29. No abstract available. PMID 32299780
- [Background] Reynolds HR, Adhikari S, Pulgarin C, Troxel AB, Iturrate E, Johnson SB, Hausvater A, Newman JD, Berger JS, Bangalore S, Katz SD, Fishman GI, Kunichoff D, Chen Y, Ogedegbe G, Hochman JS. Renin-Angiotensin-Aldosterone System Inhibitors and Risk of Covid-19. N Engl J Med. 2020 Jun 18;382(25):2441-2448. doi: 10.1056/NEJMoa2008975. Epub 2020 May 1. PMID 32356628